CLINICAL TRIAL: NCT06735560
Title: Prospective Pilot Study Assessing Imaging Performance of 89Zirconium-labelled Girentuximab (89Zr-TLX250) PET-CT in Patients With HepatoCellular Carcinoma, IntraHepatic CholangioCarcinoma or Gastro-Entero-Pancreatic Neuroendocrine Neoplasms
Brief Title: Study Assessing PET Imaging With Zirconium-labelled Girentuximab in Patients With HCC, ICC or NEN
Acronym: ELEGANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC23_0453
Record Dates: First submitted 2024-12-09; First posted 2024-12-16 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma (HCC); Intrahepatic Cholangiocarcinoma (Icc); Neuroendocrine Tumors
Keywords: immunoPET; CAIX; GEP-NEN; ICC; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension; Neuroendocrine Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 89Zr-TLX250 (Experimental): Patients will be injected with a single dose of 89Zr-TLX250.
  Interventions: Radiation: 89Zr-TLX250 PET/CT

INTERVENTIONS:
Radiation: 89Zr-TLX250 PET/CT — Patients will receive 89Zr-TLX250 for detection of CAIX-expressing tumor by PET imaging.

SUMMARY:
Precision medicine represents a major goal in oncology. It has its underpinning in the identification of biomarkers with diagnostic, prognostic, or predictive values. Gastro-entero-pancreatic neuroendocrine neoplasia (GEP-NENs) are rare tumors, but their frequency is increasing. In this context, the tumor expression of carbonic anhydrase IX (CAIX), complemented by a restricted profile in normal tissues, provides an opportunity for therapeutic targeting and precision medicine. Indeed, radiolabeling the anti-CAIX monoclonal antibody girentuximab with Zirconium 89 has shown promise as a novel positron emission tomography (PET) tracer and labeling with 177 Lutetium promise as a therapeutic agent in clear cell renal cell carcinoma (ccRCC) in the context of a theranostic approach. The purpose of this study is to evaluate the use of 89Zr-labeled girentuximab (89Zr-TLX250) as a novel, carbonic anhydrase IX (CAIX) targeted PET/CT tracer for the imaging of Gastro-Entero-Pancreatic Neuroendocrine Neoplasms, Hepatocellular Carcinoma or IntraHepatic Cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Provided written informed consent.
2. Patients aged ≥ 18 years.
3. - For basket 1 and 2: HCC or ICC histologically proven: newly diagnosed patients or patients with suspected refractory, residual, or recurrent disease.

   - For basket 3: GEP-NENs (2019 WHO classification), functioning or non-functioning, for the staging of patients with no, low or heterogeneous SSTR2 expression (who may be considered not eligible for PRRT with radiolabelled so- matostatin analogs).
4. Presence of at least one morphological evaluable lesion according to RECIST 1.1 using contrast CT/MRI.
5. Patients must have an ECOG (Eastern Cooperative Oncology Group) performance status of 0 to 2.
6. For cirrhotic patients: Child-Pugh ≤ B7.
7. Patient affiliated to or beneficiary of the National Health Service.

Exclusion Criteria:

1. Known hypersensitivity to zirconium-89, to any excipient or derivative or to radiographic contrast agents.
2. Chemotherapy, extensive external beam radiation, immunotherapy, targeted therapy, or angiogenesis inhibitors within 2 weeks prior to inclusion.
3. Radionucleide targeted therapy prior to inclusion within 6 months prior to inclusion.
4. Radioembolization within 3 months prior to inclusion.
5. Uncontrolled brain or spinal cord metastasis. Patients with a history of brain metastases must have a head CT or MRI with contrast to document stable brain disease 3 months prior to inclusion in the study.
6. Cardiac disease with New York Heart Association classification of III or IV.
7. Life expectancy shorter than 4 months.
8. Any major surgery within 4 weeks before enrollment.
9. Any uncontrolled significant medical, psychiatric or surgical condition (active infection (subjects with known human immunodeficiency virus (HIV) positive)), unstable angina pectoris, cardiac arrhythmia, poorly controlled hypertension, poorly controlled diabetes mellitus (glycated haemoglobin (HbA1c) ≥9%), uncontrolled congestive heart disease, etc.) or laboratory findings that, in the opinion of the investigator, might jeopardise the subject's safety or that would limit compliance with the objectives and assessments of the study.
10. Other known malignancies (except for fully-resected non-melanoma skin cancer or cervical cancer in situ) unless definitively treated and proven no evidence of recurrence for 2 years.
11. Women who are pregnant or breastfeeding. A serum pregnancy test will be performed at the start of the study for all female subjects of childbearing potential.
12. Patient under guardianship or trusteeship.
13. Patient under judicial protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2027-05-04 (Estimated); Study Completion 2027-08-04 (Estimated)

PRIMARY OUTCOMES:
Tumor targeting of 89Zr-TLX250 PET | Day 5
  Number of tumor lesions detected by 89Zr-TLX250 PET in comparison with the lesions identified by morphological imaging at baseline.
Tumor targeting of 89Zr-TLX250 PET | Day 5
  Location of tumor lesions detected by 89Zr-TLX250 PET in comparison with the lesions identified by morphological imaging at baseline.

SECONDARY OUTCOMES:
Evaluation of tolerability | Hour 2
  Unexpected immediate adverse events up to post-administration of 89Zr-TLX250.
Evaluation of tolerability | Day 8
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Diagnostic efficacy | Month 3
  Sensitivity of 89Zr-TLX250 PET/CT in the detection of tumor lesions as compared to a composite truth standard (determined on the basis of histology and conventional morphological or PET imaging).
Diagnostic efficacy | Month 3
  Concordance of 89Zr-TLX250 PET/CT in the detection of tumor lesions as compared to a composite truth standard (determined on the basis of histology and conventional morphological or PET imaging).
Assessment of tumor uptake | Day 8
  Tumor quantitative measures on 89Zr-TLX250 PET.
Correlation with CAIX | Day 8
  Assessment of the correlation between the normalized uptake values (SUVmax) of 89Zr-TLX250 positive lesions and CAIX histological expression will be done by comparing the 89Zr-TLX250 semi-quantitative data with the immunohistochemical results (IHC) of biopsied lesions.
Assessment of the absorbed doses | Day 0
  Quantitative biodistribution of 89Zr-TLX250 will be evaluated from sequential whole body PET-CT imaging and pharmacokinetic data.
Assessment of the absorbed doses | Day 1
  Quantitative biodistribution of 89Zr-TLX250 will be evaluated from sequential whole body PET-CT imaging and pharmacokinetic data.
Assessment of the absorbed doses | Day 5
  Quantitative biodistribution of 89Zr-TLX250 will be evaluated from sequential whole body PET-CT imaging and pharmacokinetic data.
Assessment of the absorbed doses | Day 7
  Quantitative biodistribution of 89Zr-TLX250 will be evaluated from sequential whole body PET-CT imaging and pharmacokinetic data.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Nantes, Nantes
  - AP-HP - Site de Beaujon, Paris

IPD SHARING:
Plan to Share IPD: Undecided